CLINICAL TRIAL: NCT06785337
Title: "The Effect of Inhaled Nitroglycerin on Improving Respiratory Failure in COPD Patients Admitted to Adult Intensive Care Unit"
Brief Title: "The Effect of Inhaled Nitroglycerin for COPD Patients
Acronym: iNGCOPD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Asia Said Toukhy, assistant lecturer in clinical pharmacy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-H-PhBSU-24020
Record Dates: First submitted 2025-01-06; First posted 2025-01-21 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-11

CONDITIONS: COPD; COPD III/IV
Keywords: Inhaled; nitroglycerin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (No Intervention): will receive standard COPD exacerbation treatment protocol including antibiotics, corticosteroids and bronchodilator only
- Intervention group (Experimental): will receive inhaled nitroglycerin in addition to standard COPD exacerbation treatment protocol
  Interventions: Drug: Inhaled nitroglycerin

INTERVENTIONS:
Drug: Inhaled nitroglycerin — Inhaled nitroglycerin
  Arms: Intervention group

SUMMARY:
this study aims to investigative the benefits of using nebulized nitroglycerin in improving respiratory functions in patients of late stage COPD

DETAILED DESCRIPTION:
the inhaled nitroglycerin is expected to make vasodilatation of the pulmonary arteries and arterioles which are constricted in late stages of COBD leading to ventilation/perfusion mismatching and further aggravating COPD. it will also help in delivering better antibiotic concentrations to the alveoli which help in better control of infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient's ≥ 18 years old COPD exacerbation with respiratory failure and Echo evidenced presence of pulmonary hypertension (defined as mean pulmonary artery pressure > 20 mmHg)

Exclusion Criteria:

* Profound left ventricular failure, as the decrease in pulmonary vascular resistance results in an increase in left ventricular preload. This may worsen cardiogenic pulmonary edema.
* Pregnant female patients
* Patient with hypersensitivity to nitroglycerin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary functions | 5 days after start of nebulized nitroglycerin
  Change in pulmonary functions Defined as:
  * Reduction of PaCO2 in arterial blood gases from admission value.
  * increase in Pao2 from admission value.

SECONDARY OUTCOMES:
Number of days on mechanical ventilation | 5 days after start of nebulized nitroglycerin
Dose of vasopressor therapy | 5 days after start of nebulized nitroglycerin
Reduction of WBC count | 10 days after start of nebulized nitroglycerin
Mortality rate | 10 days after start of nebulized nitroglycerin

CONTACTS AND LOCATIONS:
Locations (1):
- Haram Hospital, Haram, Giza Governorate, Egypt

REFERENCES:
- [Background] Karfunkle B, Gill J, Shirey S, Gordon R. COVID-19 Acute Respiratory Distress Syndrome and Pulmonary Embolism: A Case Report of Nebulized Nitroglycerin and Systemic Thrombolysis For Right Ventricular Failure. J Emerg Med. 2021 Nov;61(5):e103-e107. doi: 10.1016/j.jemermed.2021.07.014. Epub 2021 Jul 9. PMID 34479748
- [Background] Daunaria DK, Singh GK, Agarwal A, Mishra P. COVID-19-associated acute respiratory distress syndrome (C-ARDS): Inhaled nitroglycerin could be an efficient pulmonary vasodilator. Indian J Anaesth. 2023 Apr;67(4):403-405. doi: 10.4103/ija.ija_635_22. Epub 2023 Apr 10. No abstract available. PMID 37303880
- [Background] Daxon BT, Lark E, Matzek LJ, Fields AR, Haselton KJ. Nebulized Nitroglycerin for Coronavirus Disease 2019-Associated Acute Respiratory Distress Syndrome: A Case Report. A A Pract. 2021 Feb 5;15(2):e01376. doi: 10.1213/XAA.0000000000001376. PMID 33560642
- [Background] Mandal B, Kapoor PM, Chowdhury U, Kiran U, Choudhury M. Acute hemodynamic effects of inhaled nitroglycerine, intravenous nitroglycerine, and their combination with intravenous dobutamine in patients with secondary pulmonary hypertension. Ann Card Anaesth. 2010 May-Aug;13(2):138-44. doi: 10.4103/0971-9784.62946. PMID 20442544
- [Background] Cai YM, Zhang YD, Yang L. NO donors and NO delivery methods for controlling biofilms in chronic lung infections. Appl Microbiol Biotechnol. 2021 May;105(10):3931-3954. doi: 10.1007/s00253-021-11274-2. Epub 2021 May 3. PMID 33937932
- [Background] Polzin A, Curtis ED, Rupe E, Sang HI. Inhaled Nitroglycerin for Pulmonary Edema in Air Medical Services: A Retrospective Pilot Study. Air Med J. 2024 Mar-Apr;43(2):151-156. doi: 10.1016/j.amj.2023.11.009. Epub 2023 Dec 19. PMID 38490779
- [Background] Kline JA, Hall CL, Jones AE, Puskarich MA, Mastouri RA, Lahm T. Randomized trial of inhaled nitric oxide to treat acute pulmonary embolism: The iNOPE trial. Am Heart J. 2017 Apr;186:100-110. doi: 10.1016/j.ahj.2017.01.011. Epub 2017 Jan 27. PMID 28454823
- [Background] Monsalve-Naharro JA, Domingo-Chiva E, Garcia Castillo S, Cuesta-Montero P, Jimenez-Vizuete JM. Inhaled nitric oxide in adult patients with acute respiratory distress syndrome. Farm Hosp. 2017 Mar 1;41(2):292-312. doi: 10.7399/fh.2017.41.2.10533. PMID 28236803